CLINICAL TRIAL: NCT03843268
Title: Multi-center, Double-blind, Cross-over Randomized Study on the Use of the Medical Device "Gondola" for Motor Rehabilitation in Patients With Parkinson's Disease
Brief Title: Study on the Device "Gondola" for Motor Rehabilitation in Parkinson's Disease
Acronym: GondoPark V2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: RP 13/17
Record Dates: First submitted 2019-02-12; First posted 2019-02-18 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Automated Mechanical Peripheral Stimulation (AMPS); Gait Disorders
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in 2 groups, one starting with AMPS treatment, the other with placebo treatment. At the end of the first cycle of 6 stimulations over a 3 weeks' time (AMPS or Sham), all subject will undergo a washout period of minimum 6 weeks, then will undergo another equivalent treatment cycle (Sham or AMPS)
Who Masked: Participant, Investigator
Masking Description: Trained professionals, not directly involved in the research treatment and blind to patients group allocation, will perform clinical assessments. All subjects will undergo inpatient rehabilitation consisting of a treatment cycles using the Gondola device, once effective (AMPS treatment) and once placebo (Sham treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMPS Gondola (Active Comparator): Gondola is a portable device that runs on batteries and is fitted on both patient's feet when the patient is lying down. The device has been designed for the stimulation of two areas of both feet (first toe and metatarsal) through mechanical impulses set up for pressure, duration and sequence (Automated Mechanical Peripheral Stimulation - AMPS)
  Interventions: Device: AMPS Gondola; Device: Sham Gondola
- Sham Gondola (Placebo Comparator): The Sham treatment consist in the stimulation of the same areas through mechanical impulses different for pressure since attached to the steel stick point is positioned a rigid plastic circle with a diameter (12mm); thanks to this the induced pressure ishence lower and the surface contact bigger.
  Interventions: Device: AMPS Gondola; Device: Sham Gondola

INTERVENTIONS:
Device: AMPS Gondola — Gondola is a portable device that runs on batteries and is fitted on both patient's feet when the patient is lying down. The device has been designed for the stimulation of two areas of both feet (first toe and metatarsal) through mechanical impulses set up for pressure, duration and sequence (Automated Mechanical Peripheral Stimulation - AMPS); the treatment requires less than 2 minutes.
Device: Sham Gondola — The Sham treatment consist in the stimulation of the same areas through mechanical impulses different for pressure since attached to the steel stick point is positioned a rigid plastic circle with a diameter (12mm); thanks to this the induced pressure ishence lower and the surface contact bigger

SUMMARY:
The purpose of this research study is to evaluate safety and effectiveness of the Automated Mechanical Peripheral Stimulation (AMPS) therapy given via the Gondola™ device to improving Gait and Gait Related Disorders in patients with Parkinson'disease (PD). Gondola® is a portable device that runs on batteries and is fitted on both patient's feet when the patient is lying down. The device has been designed for the stimulation of two areas of both feet (first toe and metatarsal) through mechanical impulses set up for pressure, duration and sequence (Automated Mechanical Peripheral Stimulation - AMPS); the therapy requires less than 2 minutes.

DETAILED DESCRIPTION:
The proposed project, through a randomized multicentric, placebo controlled double-blind crossover trial aimed at evaluating the effectiveness of AMPS Gondola therapy versus Sham Gondola therapy in PD subjects. 132 in/outpatients with PD will be recruited. Subjects will be randomized in 2 groups, one starting with AMPS treatment, the other with placebo treatment. At the end of the first cycle of 6 stimulations over a 3 weeks' time (AMPS or Sham), all subjects will undergo a washout period of minimum 6 weeks, then will undergo another equivalent treatment cycle (Sham or AMPS); a follow up valuation 14 days after the end of each treatment cycle will be performed.

This project is aimed at studying and documenting the effects of the AMPS treatment given to PD patients via the Gondola device in:

1. Improving gait, reducing bradykinesia, treating Freezing of Gait symptom;
2. Improving UPDRS II and III scores;
3. Improving balance. Another goal of the study is to document the safety of the Gondola device.

ELIGIBILITY:
Inclusion criteria:

* Patients with clinically chronic and stable PD, confirmed according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnosis Criteria (UKPDSBBC);
* Age 45 and older;
* Hoehn & Yahr (H&Y) stage equal or higher than 2 in ON state;
* Ability to walk autonomously or with minimal assistance for a 10 meters' distance in OFF state;
* Antiparkinsonian treatment at a stable and optimized daily dosage during the 4 weeks prior to the study.

Exclusion criteria

* Any advanced, severe or unstable disease other than PD, which may interfere with the primary and secondary study outcome evaluations (autonomic dysfunction, diabetes, renal or hepatic failure, neoplasia, balance and gait problems of other origin).
* Cognitive impairment with MoCA < 18
* Any peripheral neurological or musculoskeletal conditions that may alter balance and/or gait.
* Severe lower limb injuries in the previous 6 months.
* History of neurosurgery or orthopedic surgery.
* History of epilepsy.
* Any drug treatment not intended to treat PD that may alter cognitive and/or motor performance.
* History of depression or other psychiatric disorders.
* Severe obesity defined as a BMI greater than 35.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Difference between effective treatment phase versus placebo treatment phase in the change of gait speed from PRE-treatment cycle to POST treatment cycle | through study completion, an average of 16 weeks
  Study success will be defined by an:
  improvement in gait speed of no less than 0,06 m/s as follows: H0: DT treatment phase - DT Sham phase < 0.06m/s v.s. Ha: DT treatment phase - DT Sham phase ≥ 0.06m/s
  Where:
  DT = VPost6 - VPre VPost 6= gait speed after 6 treatment stimulations (at the end of the treatment cycle) Vpre = gait speed before the 1st treatment stimulation (at the beginning of the treatment cycle)

SECONDARY OUTCOMES:
Change in clinical evaluation in MDS-UPDRS | through study completion, an average of 16 weeks
  Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease (MDS-UPDRS) range from 0 - less affect - to 272 - more affect
Change in clinical evaluation of step speed | through study completion, an average of 16 weeks
  step length measured in meters per second
Change in time in walking | through study completion, an average of 16 weeks
  time needed to perform the 10 meters walking test (seconds)
Change in clinical evaluation in FOG-Q | through study completion, an average of 16 weeks
  FOG-Q is a questionnaire to assess Freezing of gait (FOG) and walking among patients with Parkinson's disase (range from 0 - less affect - to 24 -more affect)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Stocchi, MD. PhD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Semprini R, Sale P, Foti C, Fini M, Franceschini M. Gait impairment in neurological disorders: a new technological approach. Funct Neurol. 2009 Oct-Dec;24(4):179-83. PMID 20412722
- [Background] Nieuwboer A, Dom R, De Weerdt W, Desloovere K, Fieuws S, Broens-Kaucsik E. Abnormalities of the spatiotemporal characteristics of gait at the onset of freezing in Parkinson's disease. Mov Disord. 2001 Nov;16(6):1066-75. doi: 10.1002/mds.1206. PMID 11748737
- [Result] Lo AC, Chang VC, Gianfrancesco MA, Friedman JH, Patterson TS, Benedicto DF. Reduction of freezing of gait in Parkinson's disease by repetitive robot-assisted treadmill training: a pilot study. J Neuroeng Rehabil. 2010 Oct 14;7:51. doi: 10.1186/1743-0003-7-51. PMID 20946640
- [Derived] De Pandis MF, Tomino C, Proietti S, Rotondo R, Gaglione M, Casali M, Corbo M, di Biase L, Galli M, Goffredo M, Stocchi F. Mechanical peripheral stimulation for the treatment of gait disorders in patients with Parkinson's disease: a multi-centre, double-blind, crossover randomized controlled trial. J Neuroeng Rehabil. 2025 Apr 8;22(1):77. doi: 10.1186/s12984-025-01574-3. PMID 40200338